CLINICAL TRIAL: NCT02847156
Title: Clinical and Microbiological Impact of Respiratory Viral Infections in the Short and Medium Term in Infants (<24 Months) With Cystic Fibrosis.
Brief Title: Impact of Respiratory Viral Infections in Infants With Cystic Fibrosis.
Acronym: PREVIMUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 69HCL14_0276
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Cystic Fibrosis; Respiratory Viral Infection
Keywords: cystic fibrosis; viruses; respiratory viral infection; children
MeSH Terms: conditions — Cystic Fibrosis; Virus Diseases | interventions — Restraint, Physical

ARMS (1):
- cystic fibrosis infants (Other): 1 year follow-up in CF infants
  Interventions: Other: Physical assessment

INTERVENTIONS:
Other: Physical assessment — 1 year follow-up in CF infants with clinical, microbiological and therapeutic assessments

SUMMARY:
Respiratory Viral Infections (RVI) are particularly frequent in young children. Old data mention the deleterious role of some viruses such as the Respiratory Syncytial Virus in young children with cystic fibrosis (CF). However, recent epidemiological data on RVI in CF children are rare and the impact of most frequent viruses such as human rhinoviruses is usually not correctly evaluated.

The aim of this study is to assess the frequency of lower and upper RVI during a 1 year follow-up in CF infants and to evaluate the impact of RVI at a clinical, microbiological and therapeutic level.

Our hypothesis is that frequent and/or clinically severe RVIs have the worst impact in the short term and without any particular link with a specific virus as previously described.

ELIGIBILITY:
Inclusion Criteria:

- infant <24 months with cystic fibrosis

Exclusion Criteria:

- patient >24 months

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of Respiratory Viral Infection | up to 12 months

SECONDARY OUTCOMES:
Identification of respiratory viruses in throat-swabs | up to 12 months
  A panel of 10 viruses will be tested using polymerase chain reaction (PCR) and RT-PCR technology.
Number of antibiotics treatments (oral or IV) | up to 12 months
Number of bronchodilator administrations | up to 12 months
Number of corticosteroids administrations | up to 12 months
Number of hospitalization or hospital admission due to upper or lower RVI | up to 12 months
Identification of bacterial flora in throat-swabs | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie VRIELYNCK, MD, Principal Investigator — Cystic Fibrosis Pediatric Reference Centrer, Hospices Civils de Lyon, 69677 Bron Cedex, France
Locations (1):
- Cystic Fibrosis Pediatric Reference Centrer, Hospices Civils de Lyon, Bron, France